CLINICAL TRIAL: NCT04865120
Title: A Monocenter, Double-blind, Comparative, Controlled, Randomized Study to Evaluate the Effect of E212657 Compared to Placebo on Long UVA Induced Pigmentation in Healthy Volunteers.
Brief Title: Photoprotection Efficacy With Sunscreen Formulas Containing the Cyclic Merocyanine Long-UVA Absorber MCE Under Long-UVA Exposure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACR_LUVA_1311
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Sunscreen Sensitivity; Ultraviolet-Induced Change in Normal Skin
Keywords: Ultraviolet A; pigmentation

STUDY DESIGN:
Intervention Model Description: Randomized double-blind mini-zones on volunteers back
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- merocyanine (Active Comparator)
  Interventions: Other: cream cyclic merocyanine
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: cream cyclic merocyanine — cream long-UVA absorber
  Arms: merocyanine
Other: placebo — placebo
  Arms: placebo

SUMMARY:
To evaluate the photo-protector effect of BC_3 (E212657) formulated in SPF compared to SPF alone on long-UVA induced pigmentation in healthy volunteers.

DETAILED DESCRIPTION:
The sun emits numerous radiations, of which 10% are constituted by ultraviolet light. Only ultraviolet B (UVB, 280-320 nm) and ultraviolet A (UVA, 320-400 nm) reach the surface of the earth. Poor penetrating UVB reach only to the deepest layers of the epidermis and cause DNA damage. UVA rays pass through the epidermis and reach the dermis due to their greater penetration property. UVA mainly generate intracellular oxidative stress. We can distinguish short UVA (320-340 nm) and long UVA (340-400 nm).

Sun exposure causes short-term consequences such as sunburn and reflects a reaction erythema, inflammatory type, and stimulation of pigmentation. One of the long-term deleterious consequences is represented by the development of skin cancers, which are the most dramatic result of sun exposure and are associated with mutations resulting from DNA damage badly repaired. The other long-term consequence is illustrated by the clinical signs of photoaging, associated with a major disruption in the dermal structure, linked both the decrease in collagen content and an increase in its degradation by some enzymes in the family of MMPs (matrix metalloproteinases). At the cellular and molecular level, many genes have their basal expression modulated in response to UV exposure (transcription factors and genes involved in DNA repair, inflammation, apoptosis, cell adhesion). Chronic sun exposure is also associated with the development or aggravation of pigmentary disorders, zones of hypo- or hyperpigmentation, actinic lentigo, melasma.

To protect ourselves from harmful effects of sun exposure, solar formulas applied to the skin, constitute a "barrier" against UV radiation. Currently, the most efficient sunscreen formulas from the market can absorb very efficiently and most of UVB and UVA rays. However, a part of long UVA (370-400nm) is not absorbed by these formulas, while these wavelengths seem to be involved in the generation of adverse biological effects on the skin, which may participate in clinical consequences of sun exposure, such as photo-aging and carcinogenesis. Biologically these wavelengths have been found to induce alteration at the tissue level, in particular the dermal layer, but also at the cellular and molecular levels, with for example the generation of oxidative stress and DNA damage.

Internal in vitro studies on skin cells in culture or on reconstructed skin showed that long UVA were the generators of oxidative stress, damage to DNA, cytotoxicity and modulation of genes or proteins involved in inflammation, the response to oxidative stress or photo-aging.

New sunscreens that are able to absorb beyond 370 nm, are now available. We have shown in an in vitro cultured cells or reconstructed skin that adding this type of filter in a state of the art formulation, allowed to shift the absorption spectrum beyond 370 nm and more. Thus it is possible to significantly reduce the biological impact of UVA long. These in vitro results strongly suggest a gain of biological protection by shifting the spectrum absorption beyond 370 nm.

The purpose of this clinical proof of concept study is to demonstrate that the addition of the Merocyanine BC_3 (E212657), a new long UVA filter, in a reference formula improves protection against a long UVA exposure in vivo in human. Safety studies have demonstrated that BC_3 (E212657) is a safe product (Non phototoxic, non irritant, non sensitizer, non photosensitizer and non Genotoxic). In vitro studies have shown versus reference a photo-protector effect on fibroblast, MMP1 and Cytokines after an 60J/cm² exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female or male volunteer;
* from 18 to 40 years old;
* uniform skin color all over on the investigational zones;
* skin type III or IV according to the Fitzpatrick classification;
* ITA° between 10° and 35° at screening visit with an authorize delta of ± 2° at inclusion visit (D1) (Individual Typologic Angle calculated value);
* female of childbearing age using a reliable mean of contraception (for at least three month before the beginning of the study, and throughout the study);
* informed about the study objectives and procedures, and able to understand them;
* willing and able to fulfill the study requirements and schedule.
* All subjects will have to give their written informed consent.

Exclusion Criteria:

* Female in pregnancy (positive pregnancy-test performed before inclusion) or lactation or without effective contraception ;
* having planned U.V. exposure of the investigational zones (sunlight or sunbeds) throughout the study;
* having used sunbed or sun exposure of the investigational zones within the 3 months before inclusion;
* having sunburn (erythema) on the back;
* dermatological disorders affecting the investigational zones (presence of naevi, freckles, excess hair or uneven skin tones, vitiligo, photo-dermatological problems);
* history of skin cancer;
* history of abnormal response to sun;
* presence of recent suntan (according to Investigator opinion) or photo-test marks;
* history of allergy, hypersensitivity, or any serious reaction to any cosmetic product;
* any concomitant medical condition that may interfere with the study conduct in the opinion of the investigator;
* having used within the month before inclusion any systemic medication for more than 5 consecutive days (e.g. steroidal and non-steroidal anti-inflammatory drugs, insulin, antihistamines, antihypertensive, antibiotics -e.g. quinolone, tetracycline, thiazides, fluoroquinolones-), or any medication known to cause abnormal responses to U.V. exposure (e.g. vitamin A derivatives, psoralen, aminolevulinic acid derivatives, etc.), or having planned to use these medications during the study;
* having used within the 3 months before inclusion any depigmenting / whitening or propigmenting topical treatments, or any systemic treatment that would interfere with the study assessments (antiinflammatory drugs, corticoids, retinoids, hydroquinone, etc.);
* unable to be contacted by phone in case of emergency;
* having participated within the 30 days before inclusion or currently participating in another clinical study.
* Deprived of liberty by adjunction or by official decision.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — from 18 to 40 years old
Enrollment: 50 (Estimated)
Dates: Start 2021-04-29 (Estimated); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Biophysical of skin color | Change from baseline at Day 7
  skin color by using Chromameter
Clinical investigator's assessment | Change from baseline at Day 7
  Visual scoring of pigmentation

SECONDARY OUTCOMES:
Recording Adverse Events, including cutaneous reactions | Change from baseline at Day 7
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP Biotechnology, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
Report final
Supporting Information: CSR